CLINICAL TRIAL: NCT00462098
Title: Randomized Controlled Trial of Hyperbaric Oxygen in Patients Who Have Taken Bisphosphonates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007527
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Osteonecrosis
Keywords: Osteonecrosis of the jaw; hyperbaric oxygen; bisphosphonates
MeSH Terms: conditions — Osteonecrosis | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HBO (Experimental): Subject receives 40 HBO sessions at 2 atmospheres of pressure over 4 weeks
  Interventions: Device: hyperbaric oxygen
- Control (Active Comparator): non-HBO comparison group
  Interventions: Device: non-treated control group

INTERVENTIONS:
Device: hyperbaric oxygen — 40 sessions of 100% oxygen at 2 atmospheres of pressure for 2 hours each
  Arms: HBO
Device: non-treated control group — no change from routine care, no HBO
  Arms: Control

SUMMARY:
Osteonecrosis of the jaw (ONJ) has recently been recognized as associated with bisphosphonate therapy, however there is little information on the natural history, treatment or prevention strategies for this condition. The purpose of this study is to determine the effectiveness of hyperbaric oxygen as a treatment. We will randomize 35 out of 70 ONJ patients to receive HBO in addition to their routine oral surgery care and follow both groups over a 2-year period.

DETAILED DESCRIPTION:
Osteonecrosis of the jaw (ONJ) has recently been recognized as associated with bisphosphonate (BP) therapy, however there is little information on the natural history, treatment or prevention strategies for this condition1. Bisphosphonates, particularly compounds containing an aliphatic chain with an amino group in the R2 position, (pamidronate, alendronate and zoledronate) are extremely effective and widely used in the treatment of breast cancer, prostate cancer, multiple myeloma and non-malignant bone disease. Although ONJ appears to develop in less than one percent of patients taking these drugs, the seriousness of the disease plus the current lack of treatment options makes this a very difficult clinical problem This study will randomize 35 out of 70 patients to receive HBO in addition to their routine oral surgery therapy for ONJ and follow both groups over a 2-year period. The study design is an interventional, prospective, randomized trial with a 2-year follow up period. Seventy subjects meeting the inclusion criteria for ONJ will be recruited by participating physicians and randomized to receive 40 HBO treatments over a 4 week period or to continue their normal oral care. No subject, HBO treated or not, will be asked to change, initiate or discontinue any ongoing therapies they may be receiving from their primary care giver for ONJ or any other medical condition. The analysis will compare remission rates between the two groups while controlling for age, gender, race, previous local trauma or surgery, tumor type, diabetes, immunosuppression, bisphosphonate duration, indication (hypercalcemia), infection, corticosteroids, and thalidomide and dental hygiene. All subjects will be closely followed throughout the 24 month course of the study with weekly contacts by phone or email to log jaw pain level as well as to record any change in general medical condition. The 17 question Duke Health Profile will be used to measure quality of life indicators at 4 key points during the study.

Comparison(s): 1) clinical remission rate in patients receiving and not receiving HBO. 2) Bone turnover and molecular measures of osteoclast signaling in ONJ patients before and after HBO and relative to non-diseased controls (labs from non-diseased controls to be obtained from a companion study).

ELIGIBILITY:
Inclusion Criteria:

* Able to consent
* Meets definition of ONJ
* Has taken amino-bisphosphonates

Exclusion Criteria:

* Unable to consent
* Ineligible for HBO
* Taking protease inhibitors for HIV
* Any past history of radiation to head or neck
* Life expectancy less than 12 months
* Tobacco use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical outcome assessments. Effect of HBO as an adjunct to the routine treatment of ONJ will be evaluated by physical exam and pain scores | Weekly for pain score. All others at: 3 months 6 months 12 months 18 months

SECONDARY OUTCOMES:
Quality of life measurements by the Duke Health Profile | 3 months, 6 months, 12 months and 18 months
Laboratory measures of bone turnover | 3 months, 6 months 12 months and 18 months
Molecular indicators of osteoclast activation (RANK, RANKL, OPG, pAKt) | 3 months 6 months 12 months 18 months

CONTACTS AND LOCATIONS:
Overall Officials: John Freiberger, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Beth-Tasdogan NH, Mayer B, Hussein H, Zolk O, Peter JU. Interventions for managing medication-related osteonecrosis of the jaw. Cochrane Database Syst Rev. 2022 Jul 12;7(7):CD012432. doi: 10.1002/14651858.CD012432.pub3. PMID 35866376